CLINICAL TRIAL: NCT00854828
Title: A Multicenter Prospective Study of Quality of Life in Adult Scoliosis
Acronym: ASLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Northwestern University (Other); New York University (Other); University of Virginia (Other); University of Louisville (Other); Maryland Spine Center (Other); Hospital for Special Surgery, New York (Other); University Health Network, Toronto (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR055176-01A2 (NIH); R01AR055176 (NIH)
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Scoliosis
Keywords: Symptomatic 40-80 y/o w/lumbar Cobb of 30 degrees; All Participants must be reasonable surgical candidate at enrollment
MeSH Terms: conditions — Scoliosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: There were 2 cohorts: Randomized and Observational, each with an operative and non-operative arm.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Intervention (Active Comparator)
  Interventions: Procedure: Surgical intervention
- Non-Operative Intervention (Active Comparator)
  Interventions: Other: Non-operative intervention

INTERVENTIONS:
Procedure: Surgical intervention — Surgical intervention as appropriate for adults with symptomatic lumbar scoliosis
  Arms: Surgical Intervention
Other: Non-operative intervention — Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc.
  Arms: Non-Operative Intervention

SUMMARY:
This is a multicenter study evaluating the effectiveness of nonoperative and operative treatments. The investigators wish to identify important clinical and radiographic determinants of outcomes in the management of adults with symptomatic lumbar scoliosis (ASLS).

Note: Enrollment was complete July 2014. National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) funding ended 2/28/17. We continue to follow enrolled subjects while we seek additional funding to follow all subjects through 8 years.

DETAILED DESCRIPTION:
Specific Aim #1: Compare the outcomes of surgery and nonoperative treatment in patients aged 40 to 80 with ASLS defined as a lumbar curve with a coronal Cobb measurement ≥ 30°, and either of the following: Oswestry (ODI) score of 20 or more; or Scoliosis Research Society Quality of Life instrument (SRS-QOL) score of 4.0 or less, in the domains of pain, function and/or appearance.

Specific Aim #2: Evaluate the impact of patient factors (age, gender, socioeconomic status, education) and comorbidities [mental health, body mass index (BMI) and bone mineral density (BMD)] on adverse events and treatment outcomes for both the nonoperative and operative arms. Incorporate these variables into a prediction model to help identify those patients most likely to benefit from either a surgical or nonoperative approach

ELIGIBILITY:
Inclusion Criteria:

* aged 40 to 80 years with
* ASLS defined as lumbar curve with a coronal Cobb measurement ≥ 30°, and either of the following: Oswestry Disability Index (ODI) score ≥ 20 or SRS-QOL score ≤ 4.0 in the domains of pain, function and/or appearance.
* If assigned to surgical intervention (by randomization or patient preference), the intervention plan would include, at a minimum, the Cobb levels of the Thoracolumbar/lumbar spine.

Exclusion Criteria:

* Substantial cardiac, pulmonary, renal or metabolic disease that, in the judgment of the surgical team, would preclude performing an operative procedure without undue risk of morbidity and mortality
* Concomitant high-grade spondylolisthesis (Grade 3)
* Prior thoracic or multiple level lumbar laminectomy or decompression [single or two level lumbar decompression (e.g., herniated disc) will not be an exclusion]
* Prior thoracic or lumbar fusion
* Osteoporosis evidence by a dual-energy x-ray absorptiometry (DEXA) T-score <-3.0 at hip or lumbar spine for patients considered to be at risk (post menopausal females, males > 60 years of age, steroid dependent rheumatoid arthritics, status post organ transplantation, etc.). Patients may be randomized prior to obtaining DEXA results. Non Surgical patients may initiate non surgical treatments prior to completion of DEXA (if required) as non surgical treatments will not affect DEXA results but DEXA must be completed and results entered within 3 months of enrollment. Surgical patient must have DEXA prior to surgical intervention.
* Neuromuscular scoliosis (e.g., spinal muscular atrophy, cerebral palsy, Parkinson's Disease, post-polio syndrome, Charcot Marie Tooth disease)
* Congenital scoliosis in the lumbar spine. Congenital anomalies of the cervical or thoracic spine are acceptable.
* Spine tumor, infection or connective tissue disorder
* Cognitively impaired or unable/unwilling to comply with follow-up
* Pregnancy or planning on conceiving during time of study involvement
* Ankylosing Spondylitis
* Past history of vertebroplasty or kyphoplasty of the thoracic or lumbar spine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith H Bridwell, MD, Principal Investigator — Washington University School of Medicine; Jon Lurie, MD, Study Director — Dartmouth-Hitchcock Medical Center; Christopher Shaffrey, MD, Study Director — University of Virginia
Locations (9):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Maryland Spine Center, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New York University, New York, New York
  - Hospital for Special Surgery, New York, New York
  - University of Virginia, Charlottesville, Virginia
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Hopital du Sacre', Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith JS, Kelly MP, Yanik EL, Baldus CR, Pham V, Ben-Israel D, Lurie JD, Edwards C, Glassman SD, Lenke LG, Buchowski JM, Carreon LY, Crawford CH 3rd, Lewis SJ, Koski T, Lafage V, Gupta MC, Kim HJ, Ames CP, Bess S, Schwab FJ, Shaffrey CI, Bridwell KH. Operative vs Nonoperative Treatment for Adult Symptomatic Lumbar Scoliosis at 8-Year Follow-Up: A Nonrandomized Clinical Trial. JAMA Surg. 2025 Jun 1;160(6):634-644. doi: 10.1001/jamasurg.2025.0496. PMID 40172880
- [Derived] Dial BL, Hills JM, Smith JS, Sardi JP, Lazaro B, Shaffrey CI, Bess S, Schwab FJ, Lafage V, Lafage R, Kelly MP, Bridwell KH. The impact of lumbar alignment targets on mechanical complications after adult lumbar scoliosis surgery. Eur Spine J. 2022 Jun;31(6):1573-1582. doi: 10.1007/s00586-022-07200-3. Epub 2022 Apr 15. PMID 35428916

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Cohort/Operative Intervention; Observational Cohort/Operative Intervention: Operative intervention: Operative intervention as appropriate for adults with symptomatic lumbar scoliosis.
- Randomized Cohort/Non-Operative Intervention; Observational Cohort/Non-Operative Intervention: Non-operative intervention: Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc.
Period: Overall Study
Arm/Group | Randomized Cohort/Operative Intervention | Randomized Cohort/Non-Operative Intervention | Observational Cohort/Operative Intervention | Observational Cohort/Non-Operative Intervention
Started (Baseline enrollment data collected and completed intervention.) | 30 (6 patients crossed over to non-operative intervention.) | 33 | 112 | 111
3 Months Post Intervention | 24 (6 missed visits) | 32 (1 missed visit) | 112 (112 (100%) of patients underwent operative treatment.) | 106 (2 missed visits. 3 withdrew.)
12 Months Post Intervention | 26 (2 missed visits. 1 withdrew. 1 deceased.) | 32 (1 withdrew. 15 (45%) crossed over to operative treatment.) | 112 | 101 (4 missed visits. 6 withdrew. 6 (5%) crossed over to operative treatment.)
24 Months Post Intervention | 27 (1 missed visit. 1 withdrew. 1 deceased. 24 patients (80%) underwent surgery.) | 31 (1 missed visit. 1 withdrew. 21 (64%) crossed over to operative treatment.) | 104 (8 missed visits.) | 94 (8 missed visits. 9 withdrew. 14 (13%) crossed over to operative treatment.)
Completed | 27 | 31 | 104 | 94
Not Completed | 3 | 2 | 8 | 17
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 9
Not completed — Missed 24mo visit | 1 | 1 | 8 | 8

BASELINE CHARACTERISTICS:
Population: Symptomatic adult lumbar scoliosis patients (ages 40-80, lumbar Cobb measurement >30° and Oswestry Disability Index (ODI) >20 or Scoliosis Research Society-22 <4.0) with no prior history of scoliosis surgery from 9 North American centers were enrolled in randomized or observational cohorts to evaluate surgery versus nonoperative treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Cohort/Operative Intervention | Randomized Cohort/Non-Operative Intervention | Observational Cohort/Operative Intervention | Observational Cohort/Non-Operative Intervention | Total
Number analyzed (Participants) | 30 | 33 | 112 | 111 | 286
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [53 to 66] | 63 [57 to 69] | 59 [53 to 64] | 61 [54 to 69] | 61 [54 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 102 | 101 | 258
  Male | 4 | 4 | 10 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 29 | 31 | 106 | 104 | 270
  Unknown or Not Reported | 1 | 2 | 3 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 8 | 13
  White | 28 | 32 | 108 | 99 | 267
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 7 | 5 | 3 | 19
  United States | 26 | 26 | 107 | 108 | 267
Scoliosis Research Society (SRS) Subscore [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 1 (worst score) to 5 (best score).
  scores on a scale | 3.2 [2.7 to 3.5] | 2.9 [2.7 to 3.5] | 3.1 [2.7 to 3.5] | 3.4 [3.0 to 3.7] | 3.2 [2.8 to 3.6]
SRS Pain Domain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 1 (worst score) to 5 (best score).
  scores on a scale | 3.0 [2.6 to 3.4] | 2.8 [2.2 to 3.2] | 2.8 [2.2 to 3.3] | 3.0 [2.6 to 3.6] | 2.9 [2.4 to 3.4]
SRS Function Domain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 1 (worst score) to 5 (best score).
  scores on a scale | 3.2 [2.8 to 3.8] | 3.0 [2.8 to 3.6] | 3.2 [2.6 to 3.8] | 3.4 [3.0 to 3.8] | 3.4 [2.8 to 3.8]
SRS Self-image Domain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 1 (worst score) to 5 (best score).
  scores on a scale | 2.8 [2.3 to 3.3] | 2.8 [2.5 to 3.2] | 2.8 [2.2 to 3.3] | 3.0 [2.7 to 3.5] | 2.8 [2.5 to 3.3]
SRS Mental Health Domain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 1 (worst score) to 5 (best score).
  scores on a scale | 3.8 [3.0 to 4.4] | 4.0 [3.2 to 4.0] | 3.8 [3.2 to 4.2] | 3.8 [3.2 to 4.4] | 3.8 [3.2 to 4.2]
Oswestry Disability Index (ODI) [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 100 (worst score) to 0 (best score).
  scores on a scale | 34 [24 to 46] | 46 [28 to 54] | 37 [26 to 48] | 32 [22 to 40] | 34 [24 to 46]
Numeric Rating Scale (NRS) Back Pain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 10 (worst score) to 0 (best score).
  scores on a scale | 7 [5 to 8] | 6 [5 to 8] | 7 [5 to 8] | 5 [4 to 7] | 6 [5 to 8]
Numeric Rating Scale (NRS) Leg Pain [Median (Inter-Quartile Range); unit: scores on a scale] — Scores range from 10 (worst score) to 0 (best score).
  scores on a scale | 4.5 [1 to 8] | 5 [0 to 6] | 4 [1 to 6] | 3 [0 to 5] | 4 [1 to 6]
Short form-12 (SF-12) Mental Component Score [Median (Inter-Quartile Range); unit: Percentile] — Percentiles range from 0 to 100 with 'norm' being 50.
  Percentile | 50 [45 to 61] | 51 [46 to 57] | 52 [41 to 59] | 51 [43 to 59] | 51 [42 to 59]
SF-12 Physical Component Score [Median (Inter-Quartile Range); unit: Percentile] — Percentiles range from 0 to 100 with 'norm' being 50.
  Percentile | 34 [27 to 42] | 31 [27 to 40] | 34 [27 to 40] | 37 [29 to 44] | 35 [27 to 42]
Lumbar Cobb Angle [Median (Inter-Quartile Range); unit: Degrees] — Lumbar Cobb angle is the measurement of the scoliosis (curve in the coronal plane) measured in degrees. Normal is 0.
  Degrees | 55 [47 to 62] | 48 [37 to 63] | 57 [45 to 69] | 48 [39 to 57] | 51 [42 to 63]
Lumbar Lordosis (T12-Sacrum) [Median (Inter-Quartile Range); unit: Degrees] — Lumbar lordosis is the sagittal plane measurement of T12 to S1 in degrees. Mean for normal adults is 64 degrees +/- 10 degrees based on 'An analysis of sagittal spinal alignment in 100 asymptomatic middle and older aged volunteers' published in SPINE, Vol 20, number 12, pp 1351-1358 in 1995.
  Degrees | -32 [-56 to -22] | -38 [-47 to -20] | -38 [-49 to -28] | -45 [-55 to -32] | -40 [-53 to -27]
Sagittal balance (C7 to Sacrum plumb) [Median (Inter-Quartile Range); unit: millimeters] — Measured in mm from mid body C7 to front of plumb in sagittal plane. Negative value indicates C7 plumb falls BEHIND sacrum. Ideal would be 0mm.
  millimeters | 27 [17 to 57] | 34 [21 to 70] | 26 [11 to 56] | 33 [16 to 55] | 30 [15 to 57]
Coronal balance [Median (Inter-Quartile Range); unit: millimeters] — Measure (in mm) mid body C7 to mid Sacrum plumb in coronal plane, Values reported in absolute values. Ideal = 0mm.
  millimeters | 13 [6 to 30] | 23 [14 to 38] | 19 [9 to 35] | 14 [8 to 26] | 18 [9 to 30]
Pelvic Incidence-Lumbar Lordosis Mismatch [Median (Inter-Quartile Range); unit: Degrees] — Mathematical difference between pelvic incidence and lumbar lordosis radiographic measurements in degrees. Differences > 10 degrees correlates with worse patient reported outcomes.
  Degrees | 14 [2 to 32] | 25 [15 to 34] | 15 [5 to 30] | 13 [1 to 28] | 16 [3 to 32]
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 4 | 1 | 3 | 9
  High school diploma or GED | 7 | 5 | 26 | 38 | 76
  Technical or associate's degree | 8 | 11 | 18 | 13 | 50
  Bachelor's degree | 7 | 6 | 28 | 31 | 72
  Graduate degree | 7 | 7 | 39 | 26 | 79
Income per yer [Count of Participants; unit: Participants]
  <$20,000 | 1 | 2 | 6 | 8 | 17
  $20,000-39,999 | 1 | 5 | 11 | 14 | 31
  $40,000-74,999 | 9 | 10 | 15 | 26 | 60
  $75,000+ | 12 | 13 | 61 | 51 | 137
  Did not report | 7 | 3 | 19 | 12 | 41
Smoking history [Count of Participants; unit: Participants]
  Current smoker | 1 | 3 | 6 | 7 | 17
  Former smoker | 11 | 13 | 31 | 32 | 87
  Never | 18 | 17 | 75 | 72 | 182
Body Mass Index [Median (Inter-Quartile Range); unit: units on a scale] — Normal adult BMI is 18.5 to 24.9
  units on a scale | 28 [23 to 31] | 25 [23 to 30] | 26 [23 to 29] | 25 [22 to 30] | 26 [23 to 30]
Osteopenia/Osteoporosis [Count of Participants; unit: Participants]
  None/Does not apply | 11 | 11 | 42 | 48 | 112
  t-score -1 to -1.5 | 12 | 11 | 32 | 20 | 75
  t-score -1.6 to -2.4 | 6 | 7 | 29 | 33 | 75
  t-score -2.5 or worse (or vertebral compression fx | 1 | 4 | 9 | 10 | 24
Hypertension [Count of Participants; unit: Participants]
  No | 16 | 17 | 70 | 68 | 171
  Yes, controlled with diet/exercise | 1 | 0 | 4 | 4 | 9
  Yes, controlled w/medication | 13 | 16 | 37 | 39 | 105
  Yes, poorly controlled w/medication | 0 | 0 | 1 | 0 | 1
Diabetes [Count of Participants; unit: Participants]
  No | 29 | 29 | 108 | 106 | 272
  Yes, controlled with diet | 0 | 0 | 0 | 2 | 2
  Yes, controlled with oral hypoglycemics | 0 | 3 | 4 | 2 | 9
  Yes, insulin dependent | 1 | 1 | 0 | 1 | 3
Depression/Anxiety/Psychiatric Disorder [Count of Participants; unit: Participants] | 11 | 9 | 35 | 22 | 77
Duration of back symptoms [Median (Inter-Quartile Range); unit: Months] | 36 [0 to 80] | 96 [12 to 240] | 12 [0 to 60] | 24 [2 to 120] | 24 [0 to 102]
Duration of leg symptoms [Median (Inter-Quartile Range); unit: Months] — Length of time patient reported having Leg symptoms at time of enrollment. If no leg symptoms, patient reported 0 months.
  Months | 3 [0 to 48] | 0 [0 to 12] | 0 [0 to 12] | 0 [0 to 12] | 0 [0 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Scoliosis Research Society Quality of Life Questionnaire (SRS QOL) Subscore
Description: Change was calculated as the SRS QOL Subscore value at 2-year minus the value at Baseline for Randomized Cohort (Intent-to-Treat analysis).
  SRS QOL Subscore value range is 1 to 5, where 5 is the best score and 1 is the worst score possible.
Time Frame: Baseline, 2-year
Population: All randomized participants were included in analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Randomized Surgical Intervention: Patients consenting to randomization and assigned to Surgical intervention: Surgical intervention as appropriate for adults with symptomatic lumbar scoliosis
- Randomized Non-Operative Intervention: Patients consenting to randomization and assigned to Non-operative intervention: Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc.
Arm/Group | Randomized Surgical Intervention | Randomized Non-Operative Intervention
Number analyzed (Participants) | 30 | 33
score on a scale | 0.5 [0.3 to 0.8] | 0.5 [0.2 to 0.7]
Statistical Analysis 1: Comparison: Randomized Surgical Intervention vs Randomized Non-Operative Intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis

2. Primary Outcome: Scoliosis Research Society Quality of Life (SRS QOL) Subscore
Description: Change was calculated as the SRS QOL Subscore value at 2-year as-treated follow-up minus the value at Baseline in the Observational cohort.
  SRS QOL Subscore value range is 1 to 5, where 5 is the best score and 1 is the worst score possible.
Time Frame: Baseline, 2-year
Population: All Observational participants were included. Crossover participants provided data in both treatment arms.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Observational Cohort Surgical Intervention: Patients consenting to Observational cohort participation, electively choosing Surgical intervention: Surgical intervention as appropriate for adults with symptomatic lumbar scoliosis
- Observational Cohort Non-Operative Intervention: Patients consenting to Observational cohort participation, electively choosing Non-operative intervention: Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc.
Arm/Group | Observational Cohort Surgical Intervention | Observational Cohort Non-Operative Intervention
Number analyzed (Participants) | 125 | 111
score on a scale | 0.7 [0.6 to 0.8] | 0.1 [0 to 0.2]

3. Secondary Outcome: Oswestry Disability Index (ODI) - Randomized Cohort
Description: Change was calculated as the ODI score at 2-year minus the value at Baseline in Randomized Cohort (intent-to-treat analysis).
  ODI score range is 0 to 100, where 0 is the best score and 100 is the worst score possible.
Time Frame: Baseline, 2-year
Population: All randomized participants were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Randomized Cohort Surgical Intervention: Patients consenting to randomization and assigned to Surgical intervention: Surgical intervention as appropriate for adults with symptomatic lumbar scoliosis
- Randomized Cohort Non-Operative Intervention: Patients consenting to randomization and assigned to Non-operative intervention: Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc.
Arm/Group | Randomized Cohort Surgical Intervention | Randomized Cohort Non-Operative Intervention
Number analyzed (Participants) | 30 | 33
score on a scale | -13 [-20 to -7] | -9 [-15 to -4]

4. Secondary Outcome: Oswestry Disability Index (ODI)
Description: Change was calculated as the ODI score at 2-year as treated follow-up minus the value at baseline.
  ODI score range is 0 to 100, where 0 is the best score and 100 is the worst score possible.
Time Frame: Baseline, 2-year
Population: All observational participants were included. Crossover participants provided data in both arms.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Observational Cohort Surgical Intervention | Observational Cohort Non-Operative Intervention
Number analyzed (Participants) | 125 | 111
score on a scale | -15 [-18 to -13] | -2 [-5 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed in *each participant* from enrollment through study completion (end of funding), an average of 3.6 years. Specific amount of time for each individual is dependent upon when he/she entered the study and if/when they withdrew from the study.
Description: Serious Adverse Events (SAE) were any events that resulted in:
  Death Hospitalization (new or prolonged) - Exception was hospitalization for index spinal deformity correction surgery.
  New disability (significant or permanent) Life threatening Unexpected but Reasonably Related to the Intervention
Groups:
- Surgical Intervention-As Treated AE's Occurring While Patient Was in Surgical Arm: Surgical intervention: Surgical intervention as appropriate for adults with symptomatic lumbar scoliosis. AE's are reported in the treatment arm (surgical or non-operative) patient was in at time of AE. A total of 171 patients had surgical intervention. This number includes non operative patients who crossed over to surgical intervention. Some patients spent time and had AEs in both treatment arms.
- Non-Operative Intervention-As Treated AE's Occurring While Patient Was on Non Operative Arm: Non-operative intervention: Non operative intervention as appropriate for treatment of adults with symptomatic lumbar scoliosis such as: injections, medications, physical therapy, etc. AE's are reported in the treatment arm (surgical or non-operative) patient was in at time of AE. A total of 150 had non operative interventions.
Arm/Group | Surgical Intervention-As Treated AE's Occurring While Patient Was in Surgical Arm | Non-Operative Intervention-As Treated AE's Occurring While Patient Was on Non Operative Arm
All-Cause Mortality (participants affected / at risk) | 3/171 | 2/150
Serious Adverse Events (participants affected / at risk) | 85/171 | 41/150
Other Adverse Events (participants affected / at risk) | 128/171 | 70/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Intervention-As Treated AE's Occurring While Patient Was in Surgical Arm (N=171) | Non-Operative Intervention-As Treated AE's Occurring While Patient Was on Non Operative Arm (N=150)
Surveillance, Epidemiology and End Results (SEER) Cancers (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 11 (11) — All Surveillance, Epidemiology and End Results (SEER) cancers occurring during the study were considered an SAE
Cardiac Events (Cardiac disorders) | 4 (6) | 5 (5) — Cardiac events that met NIAMS SAE criteria
Gastrointestinal Events (Gastrointestinal disorders) | 7 (7) | 10 (14) — GI events that met NIAMS SAE definitions
Genitourinary Event (Renal and urinary disorders) | 3 (8) | 2 (2) — Genitourinary events meeting NIAMS SAE reporting criteria
Pulmonary Event (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 3 (3) — Pulmonary related events meeting NIAMS SAE reporting guidelines
Surgeries Unrelated to Adult Symptomatic Lumbar Scoliosis (General disorders) | 32 (45) | 25 (31) — Surgical events NOT related to adult scoliosis resulting new hospitalization
Miscellaneous SAE (General disorders) | 15 (17) | 4 (6) — Misc events meeting NIAMS SAE criteria. Examples: Accidental injury, Dehydration, Altered metal status, Panic Attack, C spine stenosis, septic arthritis, anaphylactic shock, Addison's disease
Adult Lumbar Scoliosis Events (Musculoskeletal and connective tissue disorders) | 32 (66) | 1 (1) — Adult Scoliosis events meeting NIAMS SAE criteria. Examples: Lumbar stenosis, revision scoliosis spine surgeries)
Circulatory Disorders (Vascular disorders) | 5 (5) | 5 (5) — Circulatory Events meeting NIAMS SAE criteria such as transient ischemic attack, cerebrovascular accident, Deep Vein Thrombosis, Pulmonary Embolism)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Intervention-As Treated AE's Occurring While Patient Was in Surgical Arm (N=171) | Non-Operative Intervention-As Treated AE's Occurring While Patient Was on Non Operative Arm (N=150)
Musculoskeletal Event (excluding spine related symptoms) (Musculoskeletal and connective tissue disorders) | 65 (86) | 43 (56)
Medication Reaction (General disorders) | 8 (9) | 6 (6)
Endocrine System Events (Endocrine disorders) | 5 (5) | 6 (6)
Gastrointestinal Event (Gastrointestinal disorders) | 16 (16) | 8 (8)
Genitourinary Events (Renal and urinary disorders) | 8 (9) | 5 (5)
Cardiac events (Cardiac disorders) | 9 (10) | 5 (6)
Circulatory Events (Vascular disorders) | 7 (7) | 5 (6)
Hypertensive events (General disorders) | 9 (9) | 3 (4)
Non SEER cancer (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) — Basal and squamous cell skin cancers
Respiratory Events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (8)
Infectious Event (non spine) (Infections and infestations) | 7 (7) | 8 (8) — Ear, sinus, lyme disease, infected bites, herpes, etc.
Psychosocial Events (Social circumstances) | 19 (21) | 11 (11)
Reproductive (Reproductive system and breast disorders) | 5 (6) | 4 (4)
Vision Events (Eye disorders) | 4 (4) | 4 (4)
Misc events (General disorders) | 13 (13) | 11 (11) — Shingles, Low B12, tinnitus, syncope, restless leg syndrome, cat bite, neuropathies d/t chemo, etc.
Cerebrospinal fluid leak (intra-op) (Surgical and medical procedures) | 13 (13) | 0 (0)
Excessive blood loss/Intraop Coagulopathy (Surgical and medical procedures) | 8 (8) | 0 (0)
Ineffective fixation/Posterior element fracture (Surgical and medical procedures) | 2 (2) | 0 (0)
Spinal implant failure (no revision) (Musculoskeletal and connective tissue disorders) | 19 (19) | 0 (0) — Spinal implant failure (rod fracture, hook/screw pull out, etc) that did not require revision surgery prior to end of funding. Those failures that were revised were considered SAE and reported under SAEs
Proximal junctional kyphosis/breakdown (No revision required) (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0) — Proximal breakdown that required revision surgery during funding is considered an SAE and reported as SAE.
Spine wound problems (Not requiring admission) (Infections and infestations) | 3 (3) | 0 (0) — Superficial and deep wound infections that did not require a hospitalization. If hospitalization was required, it was considered an SAE and is reported under SAEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-01-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT00854828/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT00854828/SAP_001.pdf